CLINICAL TRIAL: NCT05957406
Title: Acumen HPI Smart Alerts and Smart Trends to Improve Compliance With an Intra-operative Hemodynamic Management Algorithm and Reduce Renal Injury Following Major Elective Noncardiac Surgery.
Brief Title: SMART TRENDS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2023-05
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Moderate to High-risk Noncardiac Surgery

STUDY DESIGN:
Intervention Model Description: HemoSphere Advanced Monitor with Acumen Hypotension Prediction Index (HPI) software feature, and Acumen IQ sensor
Masking Description: HemoSphere ClearSight Module and Pressure Controller, and adult Acumen IQ finger cuff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SMART TRENDS - Acumen IQ Sensor (Other): Acumen HPI Smart Alerts and Smart Trends Software Feature to guide hemodynamic management in moderate-to-high-risk noncardiac surgery.
  Interventions: Device: Acumen HPI Smart Alerts and Smart Trends Software
- SMART TRENDS - Acumen IQ Cuff (Other): Acumen HPI Smart Alerts and Smart Trends Software Feature to guide hemodynamic management in moderate-to-high-risk noncardiac surgery.
  Interventions: Device: The HemoSphere advanced monitoring platform with Acumen HPI software, and Acumen IQ sensor and Acumen IQ cuff

INTERVENTIONS:
Device: Acumen HPI Smart Alerts and Smart Trends Software — Device: Acumen HPI Smart Alerts and Smart Trends Software The Acumen HPI Smart Alerts and Smart Trends Software provides the clinician with physiological insight into a patient's likelihood of trending toward a hypotensive event. The Acumen HPI Smart Alerts and Smart Trends Software suite is enabled by the minimally invasive Acumen IQ sensor.
  Arms: SMART TRENDS - Acumen IQ Sensor
Device: The HemoSphere advanced monitoring platform with Acumen HPI software, and Acumen IQ sensor and Acumen IQ cuff — Device: HemoSphere ClearSight Module and Pressure Controller, and adult Acumen IQ finger cuff
  Arms: SMART TRENDS - Acumen IQ Cuff

SUMMARY:
A multicenter, interventional, feasibility comparison with historical controls

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* ASA Physical Status ≥ 2
* Elective noncardiac surgery with expected surgery duration ≥ 3 hours and expected post-operative length of stay of ≥ 3 days
* Planned monitoring with an arterial catheter; Cohort 2: without planned arterial catheter insertion
* General anesthesia with tracheal intubation and positive pressure ventilation

Exclusion Criteria:

* Inability to comply with the study intra-operative hemodynamic management algorithm such as surgeon request for relative hypotension or fluid restriction or avoidance of vasopressors
* Planned vasopressor or inotrope infusion during surgery
* Contraindication to intra-arterial blood pressure monitoring
* Has previously participated in the SMART TRENDS study
* Serum creatine > 2.0 mg/dL (> 175 μmol/L) or CKD stage > 3A
* Scheduled for intracranial or cardiac surgery
* Patient who is known to be pregnant
* Patients on mechanical circulatory support
* Emergency surgery
* Planned beach-chair positioning

Additional Exclusion Criteria for Cohort 2 only:

* Extreme contraction of the smooth muscle in the arteries and arterioles of the lower arm and hand, such as may be present in patients with Raynaud's disease
* Finger or hand deformity that prevents proper placement of finger cuff by visual inspection
* Inability to place Acumen IQ finger cuffs due to subject anatomy, condition, or obstructive paraphernalia (such as false nails)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
HPI Smart Alert | From start to end of non-cardiac surgery
  The proportion of HPI Smart Alert prompts displayed resulting in initiation of action within 5 minutes consistent with an intra-operative hemodynamic management algorithm.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UC Davis Medical Center, Sacramento, California
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Prisma Health, Greenville, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerra-Londono CE, Hand WR, Fleming N, Davis J, Treggiari MM, Dunkman WJ, Kumar SS, Khanna AK, Yang JT, Domino KB. Hypotension prediction index smart alerts and trends to improve compliance with goal-directed hemodynamic therapy: a feasibility study. BMC Anesthesiol. 2025 Sep 30;25(1):471. doi: 10.1186/s12871-025-03336-z. PMID 41029588